CLINICAL TRIAL: NCT02921854
Title: Detection of Circulating Biomarkers of Immunogenic Cell Death After Radiotherapy and Chemotherapy: An Exploratory Study
Brief Title: Detection of Circulating Biomarkers of Immunogenic Cell Death
Acronym: ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICD
Record Dates: First submitted 2016-09-28; First posted 2016-10-03 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All included patients (Experimental): 3 times Blood withdrawal for each patient (25ml each)
  Interventions: Other: Blood withdrawal

INTERVENTIONS:
Other: Blood withdrawal — For each patient, 3 blood withdrawals of 25 ml each will take place during treatment

SUMMARY:
In this exploratory study, the investigators will investigate if markers (molecular and immunological) of ICD or anti-tumor immunity (exosomal or molecular) can be detected in the serum of patients after high-dose radiotherapy alone or concurrent cisplatin-doublet therapy and radiotherapy. For each patient: withdraw blood at three times during treatment for analysis.

DETAILED DESCRIPTION:
The main aim of anticancer therapies is to exert cytotoxic effects on cancer cells. It recently emerged that some anticancer therapeutic modalities are capable of inducing a cell death subroutine called immunogenic cell death (ICD) that can mediate specific, sustained anticancer immunity. These observations have marked the beginning of intense research into immunoadjuvant or anticancer immunity inducing "side-effects" associated with anticancer therapies.

At present, in humans, no ICD-associated predictive biomarkers have been identified, which hampers the development of immunological strategies. No published data about human biomarkers for ICD is available.

In vitro, ICD has been found to be associated with the spatiotemporally defined emission of danger signals such as surface exposed calreticulin (CRT) or heat shock protein 90 (HSP90), secreted ATP and released TLR4 agonists like HMGB1 or HSP70. Moreover, recently it has emerged that ICD may also be associated with a "viral response-like chemokine signature (VCS)" capable of acting as both 'find me' signal (for granulocytic myeloid cells) and 'keep away' signal (for immature monocytic myeloid cells) - further details of this paradigm are under investigation.

Thus, the presence of these molecular determinants of ICD can be used to monitor the host immune status and as a predictive biomarker. Examples include: danger signals as surrogate positive biomarkers (HMGB1, HSP70 and autoantibodies against CRT/HSP90); viral-response like chemokine signature as direct positive biomarkers (IFN1A, IFN1B and CXCL10>CCL2>CXCL1).

The presence of determinants of ICD can be confirmed through the strategy of following biomarkers (in non-hematological cancers):

* Cancer cell-associated pro-tumorigenic cytokines/factors IL1A, IL10, IL6, TGF-B, VEGFA, VEFGC, IDO enzyme, CXCL12, IL8
* Immune cell-associated pro-tumorigenic cytokines/chemokines/factors IL10, IDO enzyme, TGF-B, IL4, IL5, IL13, TNF, M-CSF, GM-CSF, IL26, CXCl5, CCL7
* danger signals as surrogate positive biomarkers HMGB1, HSP70 and autoantibodies against CRT/HSP90
* Cancer cell-associated viral response-like chemokine signature IFN-a, IFN-b, CXCL9, CXCL10, CXCL1 and CCL2
* Immune cell-associated anti-tumorigenic cytokines or chemokines as positive biomarkers IL1B, IL12p70, IL15, IFNG, IL22, IL23, IL17A, IL2, CCL4, CCL5, CXCL13, CCL8, CCL19, CXCL11,CCL12, CCL17, CCL23, CCL22, CCL13, CCL24, CCL1, CCL26, CXCL2, CXCL16 Moreover, the investigators will also investigate serum-associated exosomes as possible biomarkers of an efficient antitumor response. Compared to certain soluble biomarkers (which are accessible and thus more susceptible to extracellular proteases), exosomal biomarkers can exhibit a longer half-life than their soluble equivalents, due to the "protection" provided by their encompassing lipid membrane. Therefore, the investigators are also interested in exploiting exosomes as a source of antitumor response information and as novel biomarkers of therapeutic success (those mentioned above and others under investigation).

Radiotherapy has been established through various robust lines of in vitro and in vivo evaluation to be capable of inducing ICD and anticancer immune responses. As an exploratory analysis, we will integrate lipidomics into the workflow. This has already been done in multiple disease settings and NSCLC has already proven to change lipid content in a quantifiable manner. The aim of this pilot study is to investigate the hypothesis that certain biomarkers of ICD that were identified in vitro or ex vivo are detectable in patient sera following radiotherapy and/or chemotherapy. Radiotherapy alone or concurrent cisplatin-doublet and radiotherapy will be investigated. The investigator will conduct this pilot study to gather initial data to build upon in future clinical trials, as there is no in vivo data available on this topic. Results will be published and used for future grant applications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or above.
* Diagnosed with non-small cell lung cancer
* Scheduled to receive one of the following two therapeutic strategies:

  * Concurrent cisplatin-doublet chemotherapy and radiotherapy (minimal dose of 60 Gy in fractionated non-ablative doses) in patients with stage III NSCLC
  * SBRT for stage I NSCLC: 54Gy in 3 fractions, 48 Gy in 4 fractions or 60 Gy in 8 or 5 fractions
* Is able and willing to comply with all trial requirements.

Exclusion Criteria:

1. Chronic use of corticosteroids, except when used as anti-emetics for chemotherapy or inhalers
2. NSAIDs taken until 5 days before radiotherapy or during radiation (low dose Aspirin at a maximum of 160 mg/day, is allowed)
3. Active auto-immune diseases
4. Immunosuppressive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Changes of relative protein expression / derived exosomes, linked to ICD | 5 weeks (during radiotherapy)
Changes of lipid profile for plasma / plasma, linked to ICD | 5 weeks (during radiotherapy)

SECONDARY OUTCOMES:
Changes of relative protein expression, linked to Th1/Th2 subsets | 5 weeks (during radiotherapy)

OTHER OUTCOMES:
Changes of relative protein expression, linked to vascular damage | 5 weeks (during radiotherapy)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (2):
- Unuversity Hospitals Leuven, Leuven, Belgium
- MAASTRO clinic, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided